CLINICAL TRIAL: NCT02656641
Title: Using the Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder 7-Item Scale (GAD-7) as Feedback Instruments in Brief Psychotherapy
Brief Title: Using the PHQ-9 and GAD-7 as Feedback Instruments in Brief Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Immaculata University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35156
Record Dates: First submitted 2015-11-25; First posted 2016-01-15 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Depressive Symptoms; Anxiety States, Neurotic
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Clients will complete symptom and quality of life scales before their first session and before their last or tenth session, whichever occurs first. Clients will not complete any scales during other sessions.
- Continuous Client Feedback (Experimental): Clients will complete symptom and quality of life scales before their first session and before their last or tenth session, whichever occurs first. Clients will then complete symptoms scales, specifically the Patient Health Questionnaire-9 and Generalized Anxiety Disorder 7-Item Scale before each other session. The treating clinician will review and discuss their results and at the beginning of each session.
  Interventions: Behavioral: Continuous Client Feedback
- Continuous Self Feedback (Experimental): Clients will complete symptom and quality of life scales before their first session and before their last or tenth session, whichever occurs first. Clients will then complete symptoms scales, specifically the Patient Health Questionnaire-9 and Generalized Anxiety Disorder 7-Item Scale before each other session. The treating clinician will not have access to these results.
  Interventions: Behavioral: Continuous Self Feedback

INTERVENTIONS:
Behavioral: Continuous Client Feedback — Clients complete rating scales before each therapy session. The therapist then views these results and discusses treatment progress with the client during the session.
  Arms: Continuous Client Feedback
Behavioral: Continuous Self Feedback — Clients complete rating scales before each therapy session. Progress is not reviewed with the therapist.
  Arms: Continuous Self Feedback

SUMMARY:
This study will assess the effects of client feedback, using the Patient Health Questionnaire - 9 and Generalized Anxiety Disorder 7-Item Scale, on depression and anxiety in individuals undergoing brief psychotherapy. Client feedback allows therapists to monitor treatment progress in real time. Identifying an easily accessible treatment intervention, which utilizes commonly used scales, that potentially enhances the effect of brief psychotherapy and improves treatment outcomes is a valuable endeavor with clear implications for therapy practices. It is hypothesized that clients who complete these scales each session will show greater symptom improvement than clients who do not complete the scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder, Generalized Anxiety Disorder, or Adjustment Disorder

Exclusion Criteria:

* Require a higher level of care than brief psychotherapy, or have been diagnosed with an intellectual disability, personality disorder, substance use disorder, or major medical illness

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms as assessed by Patient Health Questionnaire-9 | Baseline and end of treatment up to 10 weeks
  Assesses depressive symptoms
Change in anxiety symptoms as assessed by Generalized Anxiety Disorder 7-Item Scale | Baseline and end of treatment up to 10 weeks
  Assesses anxiety symptoms

SECONDARY OUTCOMES:
World Health Organization - Quality of Life BREF Scale | Baseline and end of treatment up to 10 weeks
  Assesses domains of physical health, psychological health, social relationships, and environment
Schwartz Outcome Scale | Baseline and end of treatment up to 10 weeks
  Monitors treatment outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Krystal G Ludwig, MA, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System - Adult Bridge Program, Wilmington, Delaware, United States

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Blais MA, Lenderking WR, Baer L, deLorell A, Peets K, Leahy L, Burns C. Development and initial validation of a brief mental health outcome measure. J Pers Assess. 1999 Dec;73(3):359-73. doi: 10.1207/S15327752JPA7303_5. PMID 10689649